CLINICAL TRIAL: NCT07092670
Title: MELAFERT: Impact of Adjuvant Therapy on FERTility in Patients With Resected MELAnoma at High Risk of Relapse. A Prospective Multicenter Observational Study
Brief Title: MELAFERT: Impact of Adjuvant Therapy on FERTility in Patients With Resected MELAnoma at High Risk of Relapse.
Status: Recruiting | Type: Observational
Sponsor: Intergruppo Melanoma Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: MELAFERT
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Melanoma; Fertility
Keywords: MELANOMA; fertility; skin cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — dabrafenib; trametinib; pembrolizumab; Nivolumab; Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum antimullerian hormone (AMH), Follicle Stimulating Hormone (FSH), 5-beta oestradiol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: BRAF/MEK inhibitors
  Interventions: Drug: Dabrafenib + Trametinib
- Cohort B: Anti-PD-1
  Interventions: Drug: Pembrolizumab; Drug: Nivolumab
- Cohort C: Observation arm
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Dabrafenib + Trametinib — There is no different use in the clinical application of the drugs reported above, the study on fertility will be implemented in the women with completely resected melanoma enrolled in the study
  Groups: Cohort A
Drug: Pembrolizumab — There is no different use in the clinical application of the drugs reported above, the study on fertility will be implemented in the women with completely resected melanoma enrolled in the study
  Groups: Cohort B
Drug: Nivolumab — There is no different use in the clinical application of the drugs reported above, the study on fertility will be implemented in the women with completely resected melanoma enrolled in the study
  Groups: Cohort B
Other: Observation — Patients who will not initiate adjuvant therapy, but will undergo observation (due to refusal, comorbidities, other reasons).
  Groups: Cohort C

SUMMARY:
Melanoma survivorship in reproductive-age women is increasing due to the advent of effective therapies in the curative setting. However, while the impact on fertility and ovarian function of chemotherapy agents is well known, there is still a lack of consistent data regarding novel the Mitogen-activated protein kinase (MAP) kinase pathway inhibitors and immune-checkpoint inhibitors (ICIs) used in melanoma.

A recent study showed that a single course of anti-PD-1 (PD, Programmed cell death protein 1) or anti-CTLA-4 (Cytotoxic T-Lymphocyte Antigen 4) reduced both the number and quality of oocytes in mice through an immune-mediated mechanism. In particular, primordial follicle damage cannot be restored, leading to relevant clinical implications.

The study aims to help to determine the impact of MAP kinase pathway inhibitors and ICIs on reproductive outcomes, and whether clinicians should discuss (and in what terms) fertility preservation techniques in reproductive-age women receiving ICIs and MAP kinase pathway inhibitors in the adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II, III, IV completely resected melanoma
2. Female sex
3. Under 40 years of age
4. Not previously treated with chemotherapy and/or radiotherapy
5. Being able to give written informed consent.

Exclusion Criteria:

1. Unresectable melanoma
2. Predisposing conditions for infertility
3. Early menopause or family history of early ovarian failure (idiopathic, < 45 years)
4. Previous bilateral ovariectomy or other ovarian surgery
5. Personal history of autoimmune diseases, endocrine disorders (except for hypothyroidism)
6. Personal history of severe mental disorders associated with infertility (e.g., nervous anorexia) and/or requiring treatments that could impair fertility
7. Inability to give written informed consent.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Reproductive-age female patients with completely resected stage II, III, IV melanoma, irrespective of BRAF mutational status, with no previous history of chemo, radiation therapy and/or ovarian surgery.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2032-08 (Estimated)

PRIMARY OUTCOMES:
serum antimullerian hormone (AMH) | 18 months after the start of therapy
  To evaluate, in women of childbearing age, the variation in ovarian reserve after completion of adjuvant therapy with BRAF/MEK inhibitors or anti-PD-1 agents

SECONDARY OUTCOMES:
To assess long-term fertility preservation after completion of adjuvant therapy To assess the early impact on fertilitY preservation of a short course of therapy | • AMH at 3 months after the start of adjuvant therapy • AMH at 12 months after the start of adjuvant therapy
  correlation between baseline/post-treatment serum AMH and pregnancy rate correlation between baseline/post-treatment serum AMH and menstrual activity ratio between desired (Gd)/ obtained (Go) pregnancies other reproductive outcomes

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - Ospedale Oncologico "Giovanni Paolo II", Bari
  - IRCCS Ospedale Policlinico San Martino, Oncologia Medica 2, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero-Universitaria, Modena, Modena
  - Istituto Nazionale Tumori "Fondazione Pascale", Napoli
  - IOV Istituto Oncologico Veneto, Padua
  - Azienda Ospedaliera Santa Maria della Misericordia - Unità di Oncologia Medica., Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Università degli Studi di Siena - U.O.C. Immunoterapia Oncologica Azienda Ospedaliera Universitaria Senese, Siena
  - Università di Torino - Clinica Dermatologica, Torino

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT07092670/Prot_SAP_000.pdf